CLINICAL TRIAL: NCT00635271
Title: Identification of Biomarkers in Exhaled Breath Condensates From Asthmatic Patients
Brief Title: Biomarkers in Exhaled Breath From Asthmatic Patients
Status: Terminated | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 080081; 08-H-0081
Record Dates: First submitted 2008-03-08; First posted 2008-03-13 (Estimated); Last update posted 2019-12-05 (Actual); Status verified 2012-11-28

CONDITIONS: Asthma
Keywords: Asthma; Biomarker; Exhaled Breath Condensate; Cytokine; Healthy Volunteer; HV
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
This study will look for a relationship between asthma and factors released from the lungs in exhaled breath. If a relationship can be established, the identified factors may be used as biomarkers to predict episodes of increased asthma symptoms so that medications can be given to prevent the onset of an asthma attack.

Healthy volunteers and people who have had asthma for at least 1 year may be eligible for this study. Candidates must be between 18 and 75 years of age.

Participants undergo blood tests and breathing tests. For the latter, participants breathe into a machine before and after inhaling an asthma medication called albuterol. The machine measures the volume of air the subject can breathe out. Participants also provide a sample of exhaled breath by breathing normally for up to 30 minutes while wearing a mask devised for the procedure. Pulse rate, oxygen saturation and wheezing are monitored during the breath collection.

DETAILED DESCRIPTION:
Asthma is a major public health problem that is associated with significant morbidity and mortality. Patients at increased risk for asthma decompensations include those with severe asthma that is refractory to therapy, as well as patients with poorly controlled disease due to inadequate treatment. The aim of this exploratory specimen procurement protocol is to develop a non-invasive method for the detection of asthma-specific biomarkers in exhaled breath condensates (EBC) utilizing a novel collection device that was engineered at the Johns Hopkins University Applied Physics Laboratory. Biomarkers in EBC will be identified by mass spectroscopy. We propose that the identification of biomarkers in EBC that correlate with airway inflammation and disease activity may be used to guide therapy and prevent exacerbations in asthmatic patients.

ELIGIBILITY:
* INCLUSION CRITERIA - ASTHMA:

Patients will be between 18 and 75 years of age, male or female, with a diagnosis of asthma for at least one year.

Oxygen saturation on room air greater than or equal to 92 percent.

EXCLUSION CRITERIA - ASTHMA:

Diagnosis of a pulmonary disorder other than asthma (for example: chronic bronchitis, emphysema, cystic fibrosis, bronchiectasis, sarcoidosis, HIV-related lymphocytic airway inflammation).

Cigarette smoking within the past 3 months or a prior history of greater than 10 cumulative pack-years.

History of coronary artery disease.

INCLUSION CRITERIA HEALTHY VOLUNTEERS:

Research volunteers will be between 18 and 75 years of age, male or female.

Oxygen saturation on room air greater than or equal to 92 percent.

EXCLUSION CRITERIA HEALTHY VOLUNTEERS:

Same as the asthmatic exclusion criteria plus a history of asthma.

Reversible Airflow Obstruction (increase in FEV (1) by 12 percent and 200 cc after inhaled beta 2-agonist)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2008-02-29; Study Completion 2012-11-28

CONTACTS AND LOCATIONS:
Overall Officials: Stewart J Levine, M.D., Principal Investigator — National Heart, Lung, and Blood Institute (NHLBI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Braman SS. The global burden of asthma. Chest. 2006 Jul;130(1 Suppl):4S-12S. doi: 10.1378/chest.130.1_suppl.4S. PMID 16840363
- [Background] El-Ekiaby A, Brianas L, Skowronski ME, Coreno AJ, Galan G, Kaeberlein FJ, Seitz RE, Villaba KD, Dickey-White H, McFadden ER Jr. Impact of race on the severity of acute episodes of asthma and adrenergic responsiveness. Am J Respir Crit Care Med. 2006 Sep 1;174(5):508-13. doi: 10.1164/rccm.200603-431OC. Epub 2006 Jun 8. PMID 16763217
- [Background] Wenzel S. Severe asthma in adults. Am J Respir Crit Care Med. 2005 Jul 15;172(2):149-60. doi: 10.1164/rccm.200409-1181PP. Epub 2005 Apr 22. PMID 15849323